CLINICAL TRIAL: NCT03956537
Title: Fusion With the Neo Pedicle Screw and Cage Systems: A Post Market Clinical Follow-up Study
Brief Title: PMCF Neo Pedicle Screw and Cage Systems
Status: Active, not recruiting | Type: Observational
Sponsor: Neo Medical SA (Industry)
Collaborators: ConfinisCPM (Unknown)
Responsible Party: Sponsor
Other Study IDs: NeoPMCF01
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spinal Stenosis; Spinal Tumor; Trauma; Pseudoarthrosis of Spine
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spinal Stenosis; Spinal Cord Neoplasms; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pedicle screw system alone
  Interventions: Device: NEO Pedicle Screw System™
- Pedicle screw system with cages
  Interventions: Device: NEO Pedicle Screw System™; Device: Neo Cage System™

INTERVENTIONS:
Device: NEO Pedicle Screw System™ — The NEO Pedicle Screw System™ is intended to provide immobilization and stabilization of spinal segments in skeletally mature patients as an adjunct to fusion.
Device: Neo Cage System™ — Neo Cage System™ is intended to be used with bone graft material to facilitate interbody fusion and to be used with the NEO Pedicle Screw System™
  Groups: Pedicle screw system with cages

SUMMARY:
The objectives of this clinical observational study is to evaluate the safety and efficacy (performance) of the Neo Pedicle Screw System™ and the Neo Cage System™ interbody fusion device. To demonstrate non-inferiority of safety and function to an historical control from the published medical literature on competitive devices.

ELIGIBILITY:
Inclusion criteria:

* Patient has undergone or is intended to undergo surgery with the Neo Pedicle Screw System™, standalone or in combination with the Neo Cage System™, for any of the approved indications as defined in the respective labelling
* Patient has participated in or is willing to participate in the routine postoperative follow-up program
* Patient is willing to provide written informed consent

Exclusion criteria:

* Patient is under the age of 18 or skeletally immature
* Patient had or has a contraindication to surgery or to any of the implant systems used in the study, as defined in the respective labelling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total, approximately 150 patients will be recruited and enrolled to ensure that at least 132 patients are evaluable at 12 and 24 months. Patients are recruited consecutively, retrospectively as well as prospectively. The potential patients to be recruited have either already been implanted or are planned to be implanted with the Neo Pedicle Screw System (Arm 1) or Neo Cage System and Neo Pedicle Screw System (Arm 2).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient´s function from baseline to 12 months | 12 months
  Clinical outcome in function as measured by the 100 point Oswestry Disability Index (ODI). Zero is equated with no disability and 100 is the maximum disability possible.
The rate of cage migration in cage-plus-screw systems. | 12 months and 24 months post operatively
  Defined as posterior movement of the cage past the posterior wall of the vertebral body.
The rate of pedicle screw loosening in screw only and cage-plus-screw systems. | 12 months and 24 months post operatively
  A radiolucent zone, >1mm, surrounding the pedicle screw seen in radiograhs

CONTACTS AND LOCATIONS:
Overall Officials: David C Noriega, PhD, MD, Principal Investigator — Spine Center, University Hospital Valladolid, Valladolid, Spain; Yasser Abdalla, MD, Principal Investigator — Dep. of Neurosurgery, Nordwest Krankenhaus Sanderbusch, Sande, Germany
Locations (2):
- Dep. of Neurosurgery, Nordwest Krankenhaus Sanderbusch, Sande, Germany
- Spine Center, University Hospital Valladolid, Valladolid, Spain